CLINICAL TRIAL: NCT00214071
Title: Influence of Obstructive Sleep Apnea on Humoral and Cell-Mediated Vaccine Responses
Brief Title: Immunological Consequences of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2003-284
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2009-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza vaccine

SUMMARY:
Obstructive sleep apnea (OSA) is a medical problem whose importance is increasing in recognition and awareness. OSA is associated with the development of hypertension and other cardiovascular diseases (1,2). OSA has pathophysiologic characteristics that are known to negatively impact immune function. Both sleep deprivation and hypoxia, hallmarks of OSA, impair immune responses (6,8,11). In addition, patients with OSA are frequently obese and obesity may be associated with increased chance of infections and immune impairment (14,15). Adipose cells are known to secrete cytokines and hormones that are involved in the immune response such as leptin, tumor necrosis factor alpha and interleukin-6 (16-19). Thus, it seems very likely that OSA may impact antigen-specific immune responses. Although it is known that characteristics of OSA impact immune function, it is not known what effects clinical OSA has on immunity.

The central hypothesis of this application is that that patients with obstructive sleep apnea will have attenuated cell-mediated and humoral immune responses to influenza vaccine compared to matched control subjects. Our hypothesis has been formulated on the basis that patients with OSA are sleep deprived and experience repeated hypoxemia that negatively impact both humoral and cell-mediated immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any immunocompromising diseases or medical conditions
* Not taking any immune modifying medications or supplements
* Significant obstructive sleep apnea as verified by complete overnight polysomnography with apnea-hypopnea index (AHI) > 15 events per hour (sleep apnea subjects)
* Free of sleep disordered breathing verified by complete overnight polysomnography (AHI < 5 events per hour) or oximetry (< 5 desaturations per hour) (control subjects)

Exclusion Criteria:

* Documented history of allergy to influenza vaccine or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be mean lymphocyte interferon- ÿ (IFN- ÿ) production at 14 days (measured by ELISA)

SECONDARY OUTCOMES:
Mean influenza antibody concentrations (pre- and post-immunization) with standard deviations will be calculated and compared between sleep apnea and control patients.

CONTACTS AND LOCATIONS:
Overall Officials: John M Dopp, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States